CLINICAL TRIAL: NCT04245137
Title: A Cross-sectional Study of Female Pelvic Floor Surface Electromyography in Chinese Healthy Female
Brief Title: Reference Intervals of the sEMG of the Pelvic Floor in Healthy Female
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Xi'an People's Hospital (Xi'an Fourth Hospital) (Other); Maternal and Child Health Hospital of Anhui Province (Unknown); Ningbo Women & Children's Hospital (Other); Gansu Province Maternal and Child Care Hospital (Unknown); Foshan Maternity and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: sEMG-Normal
Record Dates: First submitted 2020-01-26; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pelvic Floor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multi-center survey of surface electromyography (sEMG) of pelvic floor muscles in healthy female. The aim of the study is to get the reference interval of normal pelvic floor sEMG from Chinese women.

DETAILED DESCRIPTION:
Pelvic floor dysfunction is a group of diseases caused by the damage of pelvic floor supporting structure. Pelvic floor muscles play an important role in the maintenance of pelvic floor function. Surface electromyography (sEMG) has been widely used to evaluate the function of pelvic floor muscles. The sEMG tests, which include pretest and posttest resting amplitude (µV), as well as phasic, tonic and endurance contractile amplitude (µV), are performed using Vishee neuro-muscle stimulator (MyoTrac Infiniti, model SA9800, Thought Technology Ltd., Montreal, Canada), following the Glazer protocols. A pear-shaped vaginal probe (serial number DYS180610, type VET-A, produced by Nanjing Vishee Medical Technology, Ltd.) is placed into the vagina when sEMG tests are performed. This is a cross-sectional survey. The reference intervals of pelvic floor sEMG in healthy female are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* a. Having sex life and tolerable to vaginal examination b. There were no symptoms related to pelvic floor dysfunction; c. The modified Oxford grading system was 4 or 5; d. No birth or 2 years after the last delivery;

Exclusion Criteria:

* a. Duration of pregnancy and lactation; b. Within 2 years after delivery; c. Acute inflammation of vagina or discomfort of vagina; d. History of pelvic floor dysfunction: leakage of urine in the past 1 month when coughing / sneezing / lifting; leakage of urine in the past 1 month when urgency fecal incontinence in the past 1 month; usually have a bulge or something falling out that can be seen or felt in vaginal area; Pain in the abdomen or lumbosacral and buttocks below the navel for more than 6 months; e. History of radical pelvic surgery (cervical cancer, rectal cancer, bladder cancer, etc.); f. History of hysterectomy and subtotal hysterectomy; g. History of pelvic floor surgery (anti-incontinence and prolapse surgery); h. History of pelvic radiotherapy; i. Nervous system diseases that significantly affect muscle function; j. Those who can't cooperate with pelvic floor contraction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: healthy females with no symptoms of pelvic floor dysfunciton and normal contraciton strength, and at least 2 yrs postpartum.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
resting amplitude (µV) pre baseline | 1 day
  pretest one minute rest

SECONDARY OUTCOMES:
coefficients of variability pre baseline | 1 day
  standard deviation divided by amplitudes at pretest resting period
maximum rapid contraction amplitude (µV) | 1 day
  five rapid contractions (Flicks) with a 10 second rest before each one (phasic).
recovery time at termination of rapid contraction(second) | 1 day
  recovery time until all muscles relax
average amplitude of tonic contraction(µV) | 1 day
  five 10 second contractions with a 10 second rest before each one (tonic)
coefficients of variability for the tonic contraction | 1 day
  standard deviation divided by amplitudes at tonic contraction period
recovery time at termination of tonic contraction(second) | 1 day
  recovery time until all muscles relax
average amplitude of endurance contraction(µV) | 1 day
  A 10 second rest followed by a single endurance contraction of 60 seconds (endurance)
coefficients of variability for the endurance contraction | 1 day
  standard deviation divided by amplitudes at endurance contraction period
resting amplitude (µV) post baseline | 1 day
  after-test one minute rest
coefficients of variability post baseline | 1 day
  standard deviation divided by amplitudes at after-test resting period

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — zhu_julie@vip.sina.com
Locations (7):
- China (7):
  - Maternal and Child Health Hospital of Anhui Province, Hefei, Anhui
  - Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Gansu Province Maternal and Child Care Hospital, Lanzhou, Gansu
  - Foshan Maternal and Child Health Care Hospital, Foshan, Guangdong
  - the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Xi'an' Fourth Hospital, Xi’an, Shanxi
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No